CLINICAL TRIAL: NCT02319629
Title: Preventive Therapy With Ursodiol to Reduce the Incidence of Gallstones Formation in Patients After Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Nasser Sakran, MD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EMC- 0129-12 -CTIL
Record Dates: First submitted 2014-12-03; First posted 2014-12-18 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Morbid Obesity
Keywords: Morbid obesity,; Cholelithiasis; Bariatric surgery; Ursodiol
MeSH Terms: conditions — Obesity, Morbid; Cholelithiasis | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- URSODIOL - URSODEOXYCHOLIC ACID (Experimental): 300 mg twice a day
  Interventions: Drug: URSODIOL
- placebo (Placebo Comparator): placebo twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: URSODIOL — preventive treatment with Ursolit to reduce the incidence of gallstones formation after bariatric surgery
  Other Names: URSODEOXYCHOLIC ACID
  Arms: URSODIOL - URSODEOXYCHOLIC ACID
Drug: Placebo
  Arms: placebo

SUMMARY:
Risk factor of cholelithiasis is rapid weight loss after bariatric surgery and change in the gallbladder function which is secondary to surgery. Many observational studies support this fact, and a high incidence of 28% -71% after gastric bypass surgery (RYGB) was reported in them. According to another publication, the incidence of gallbladder diseases is 5-36% after jejunoileal bypass surgery and 2.8-36% after gastric bypass surgery.

DETAILED DESCRIPTION:
Study format: Prospective, randomized, blinded study. 266 candidates for sleeve gastrectomy or gastric bypass surgery due to morbid obesity with BMI range of 40-50 and aged 18-65 will be studied.

The patients will be randomly divided into two groups (according to the last digit of the identity card number):

1. Treatment group will receive preventive therapy with Ursodiol 600 mg per day as of day 10 after the surgery (at the first routine visit after the surgery) and for six months or until the formation of gallstones.
2. Placebo group will receive placebo as of day 10 after the surgery (at the first routine visit after the surgery) and for six months or until the formation of gallstones.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for sleeve gastrectomy or gastric bypass surgery due to morbid obesity with BMI range of 40 to50.
* Aged 18 to 65.
* No presence of gallstones.
* Patients who have signed the consent form.

Exclusion Criteria:

* Minors,
* Pregnant women,
* Age over 65,
* Sensitive to Ursodiol,
* Gallstones,
* Biliary tract pathologies,
* Gallbladder wall thickening,
* Patients after cholecystectomy,
* Patients participating in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of gallstones formation after bariatric surgery | six month
  - Six months after the surgery the subjects will be invited to re-evaluation of the presence of gallstones using:
  1. Clinical interview: Did he experience epigastric pain? Was he hospitalized with diagnosis of biliary colic or cholecystitis?
  2. US of the upper abdomen to assess the presence of gallstones, gallbladder wall thickening or other disorder.
  3. Blood tests for liver functions and lipids profile

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Sakran, MD, Principal Investigator — Technion - Israel Institute of Technology, Faculty of Medicine
Locations (1):
- surgery department A, Afula, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Sakran N, Dar R, Assalia A, Neeman Z, Farraj M, Sherf-Dagan S, Gralnek IM, Hazzan R, Mokary SE, Nevo-Aboody H, Dola T, Kaplan U, Hershko D. The use of Ursolit for gallstone prophylaxis following bariatric surgery: a randomized-controlled trial. Updates Surg. 2020 Dec;72(4):1125-1133. doi: 10.1007/s13304-020-00850-2. Epub 2020 Jul 14. PMID 32666477